CLINICAL TRIAL: NCT05194384
Title: Eastern Siberia PCOS Epidemiology & Phenotype Study (ESPEP Study)
Brief Title: Eastern Siberia PCOS Epidemiology & Phenotype Study
Status: Completed | Type: Observational
Sponsor: Federal State Public Scientific Institution, Scientific Center for Family Health and Human Reproduction Problems (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); University of Southern California (Other); Penn State University (Other); Hacettepe University (Other); University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Larisa Suturina, The Head of the Department, Federal State Public Scientific Institution, Scientific Center for Family Health and Human Reproduction Problems
Other Study IDs: 16
Record Dates: First submitted 2022-01-04; First posted 2022-01-18 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: PCOS
Keywords: PCOS; phenotype; Eastern Siberia; Epidemiology; prevalence; hyperandrogenism; mF-G score; PCOM; unselected population
MeSH Terms: conditions — Hyperandrogenism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The investigators obtain blood for DNA extraction at the screening visit. Blood is sent to an SC FHHRP facility where DNA is extracted and stored for future analyses.

SUMMARY:
This multicenter, institution-based, cross-sectional study evaluates the prevalence of polycystic ovary syndrome (PCOS) and PCOS phenotype in Eastern Siberia - the unique region of the Russian Federation with a multi-raced population living in similar geographic and socio-economic conditions for centuries. Therefore, the investigators considered this population optimal for epidemiological research.

DETAILED DESCRIPTION:
Polycystic Ovarian Syndrome (PCOS) has a high prevalence and is a significant reproductive, metabolic, and psychosocial disorder. Several studies have demonstrated that PCOS affects from 6% (defined by NIH 1990 criteria) to 19.5% (under Rotterdam 2003 criteria) of reproductive-aged women (Jalilian et al., 2015; Bozdag et al., 2016). The prevalence of PCOS and its symptoms may vary according to geography and race/ethnicity (Huang et al., 2016; Ding et al., 2017). Clinical studies indicate variations in the presence and severity of PCOS and its clinical symptoms: hirsutism, obesity, insulin resistance by race and ethnicity. Unfortunately, there is a lack of data on the prevalence of PCOS and its phenotype in many geographic regions, in particular, in one of the largest countries in the world, Russia.

Objectives: To determine the prevalence of PCOS and the PCOS phenotypes in unselected (medically unbiased) premenopausal women in the Eastern Siberia region.

Study design and population: this is the multicenter, institution-based, cross-sectional Eastern Siberia PCOS Epidemiology & Phenotype (ESPEP) Study, conducted in Irkutsk Region and the Burjat Republic (Russia) during 2016-2019 yrs. ESPEP included premenopausal women aged 18 to 44 yrs, Caucasians, Asians, or those of mixed-race, recruited during an obligatory early medical employment assessment, and provided written informed consent. The study is approved by the Institutional Ethics Committee of the Scientific Center for Family Health a Human Reproduction (Irkutsk, Russian Federation).

Methods. Subjects are evaluated consecutively, including questionnaires, anthropometry, and vital signs, gynecological examination, modified Ferriman-Gallway (mF-G) scoring, pelvic ultrasound, and blood sampling. For PCOS diagnosis the investigators use the Rotterdam (2003) criteria. Serum samples are analyzed for total testosterone (TT) using LC-MS/MS. DHEAS, sex hormone-binding globulin (SHBG), prolactin, TSH, and 17-OHP are assessed by ELISA. Free Androgen Index (FAI) is calculated (i.e. [TT/SHBG] x 100). The upper normal limit (UNL) for the mF-G score is determined using a 2k-cluster analysis in the total study population. The upper normal limits (UNL) for TT, FAI, and DHEAS are determined from the 98th percentiles for these parameters in )women, identified as the "super-controls". Pelvic ultrasound (U/S) is performed by 3 experienced specialists with the appropriate intra/inter-observer variations, using Mindray М7 (MINDRAY, China), a transvaginal probe (5,0-8,0 МHz) or transabdominal probe (2,5-5,0 MHz). Ovarian volume is determined by the following formula: length x width x height x 0,523.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Female
* Aged 18 to 44
* All races and ethnic backgrounds

Exclusion criteria:

* Current pregnancy or lactation
* History of hysterectomy, bilateral oophorectomy, endometrial ablation, uterine artery embolization
* Current or previous (within 3 months) hormonal medications or insulin-sensitizers intake
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study
* Unwillingness to participate or difficulty understanding the consent processes or the study objectives and requirements

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: An unselected women from Eastern Siberia aged 18 to 44 years, Caucasians, Asians, or women of mixed race, recruited in Irkutsk Region and the Burjat Republic (Russia) during an obligatory early medical employment assessment in 2016-2019.
Sampling Method: Non-Probability Sample
Enrollment: 1148 (Actual)
Dates: Start 2016-04-03 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The prevalence of PCOS (overall and by race) in unselected (medically unbiased) women from Eastern Siberia ages 18 to 44 years | March 2016-December 2019
  PCOS is defined in women ages 18-44 years by the Rotterdam 2003 criteria/ Two of three features, including oligo- or anovulation (OA), clinical and/or biochemical signs of hyperandrogenism (HA), and polycystic ovarian morphology (PCOM), is required, after exclusion of related disorders.
  Exclusion of related disorders includes uncompensated thyroid dysfunction, uncompensated hyperprolactinemia and 21-hydroxylase deficient non-classic congenital adrenal hyperplasia (NC-CAH).

SECONDARY OUTCOMES:
The distribution of PCOS phenotypes among the women diagnosed with PCOS in the above objective, overall and by race. | March 2016-December 2019
  PCOS subphenotypes are defined based on the combination of clinical and biochemical PCOS features in women aged 18-44 years as follows:
  Phenotype A - clinical and/or biochemical hyperandrogenism (HA) and oligo-anovulation (OA)/menstrual dysfunction (MD), and polycystic ovarian morphology (PCOM); B - HA and OA/MD; C - HA and PCOM; and D - OA/MD and PCOM.

CONTACTS AND LOCATIONS:
Overall Officials: Larisa V Suturina, PhD, MD, Prof, Principal Investigator — Federal State Public Scientific Institution, Scientific Center for Family Health and Human Reproduction Problems. Irkutsk, Russia; Daria V Lizneva, PhD, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai, New York, NY, USA; Frank Stanczyk, PhD, Prof, Study Chair — Keck School of Medicine, University of Southern California, Los Angeles, CA, USA; Richard S Legro, MD,Prof, Study Chair — Hershey Medical Center, Penn State College of Medicine, Penn State University, Hershey, PA, USA; Bulent O Yildiz, PhD, MD, Prof, Study Chair — Hacettepe University School of Medicine, Hacettepe, Ankara, Turkey; Ricardo Azziz, PhD, MD, Prof, Study Chair — School of Public Health, University at Albany, SUNY, Albany, and School of Medicine, University of Alabama at Birmingham, Birmingham, USA
Locations (1):
- Federal State Public Scientific Institution, Scientific Center for Family Health and Human Reproduction Problems, Irkutsk, Irkutsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
For continued research, IPD data from the ESPEP study will be available to other researchers who have developed important research questions that can be answered by these valuable data. This data access policy applies to all individuals or organizations who would like to utilize data from the ESPEP Study.
  ESPEP study data may be requested by researchers from various institutions for research purposes only, by submitting an expression of interest (EoI), which should include brief information about a Project leader's name, institution, a title of the potential project, and ethical approval from the Ethics Committee, and a summary of the proposed project.
  IPD to be shared may include de-identified socio-demographic, clinical data, as well as lab tests results
Supporting Information: Study Protocol, ICF
Time Frame: The data is currently available, without time limitations
Access Criteria: Requests for access to data will be reviewed by the Sponsor and the Steering Committee of the ESPEP study A Statement of Data Use and a Confidentiality Statement must be signed by any person associated with the project including those who present results, or whose name appears on a publication that is associated with the project. Data access will not be granted until these documents are signed.
  In signing the Statement of Data Use the lead researcher acknowledges responsibility for ensuring adequate facilities and resources to enable the project to progress in a reasonable manner. Full acknowledgment of the source of data used must be provided in any publications that arise from access to and use of the data as set out in the publication policy

REFERENCES:
- [Background] Jalilian A, Kiani F, Sayehmiri F, Sayehmiri K, Khodaee Z, Akbari M. Prevalence of polycystic ovary syndrome and its associated complications in Iranian women: A meta-analysis. Iran J Reprod Med. 2015 Oct;13(10):591-604. PMID 26644787
- [Background] Bozdag G, Mumusoglu S, Zengin D, Karabulut E, Yildiz BO. The prevalence and phenotypic features of polycystic ovary syndrome: a systematic review and meta-analysis. Hum Reprod. 2016 Dec;31(12):2841-2855. doi: 10.1093/humrep/dew218. Epub 2016 Sep 22. PMID 27664216
- [Background] Huang Z, Yong EL. Ethnic differences: Is there an Asian phenotype for polycystic ovarian syndrome? Best Pract Res Clin Obstet Gynaecol. 2016 Nov;37:46-55. doi: 10.1016/j.bpobgyn.2016.04.001. Epub 2016 May 18. PMID 27289337
- [Background] Ding T, Hardiman PJ, Petersen I, Wang FF, Qu F, Baio G. The prevalence of polycystic ovary syndrome in reproductive-aged women of different ethnicity: a systematic review and meta-analysis. Oncotarget. 2017 Jul 12;8(56):96351-96358. doi: 10.18632/oncotarget.19180. eCollection 2017 Nov 10. PMID 29221211
- [Derived] Lazareva L, Suturina L, Atalyan A, Danusevich I, Nadelyaeva I, Belenkaya L, Egorova I, Ievleva K, Babaeva N, Lizneva D, Legro RS, Azziz R. Ovarian Morphology in Non-Hirsute, Normo-Androgenic, Eumenorrheic Premenopausal Women from a Multi-Ethnic Unselected Siberian Population. Diagnostics (Basel). 2024 Mar 22;14(7):673. doi: 10.3390/diagnostics14070673. PMID 38611586
- [Derived] Suturina L, Lizneva D, Atalyan A, Lazareva L, Belskikh A, Bairova T, Sholokhov L, Rashidova M, Danusevich I, Nadeliaeva I, Belenkaya L, Darzhaev Z, Sharifulin E, Belkova N, Igumnov I, Trofimova T, Khomyakova A, Ievleva K, Babaeva N, Egorova I, Salimova M, Yildiz BO, Legro RS, Stanczyk FZ, Azziz R. Establishing Normative Values to Determine the Prevalence of Biochemical Hyperandrogenism in Premenopausal Women of Different Ethnicities from Eastern Siberia. Diagnostics (Basel). 2022 Dec 22;13(1):33. doi: 10.3390/diagnostics13010033. PMID 36611327